CLINICAL TRIAL: NCT01416935
Title: Anti-Arrhythmic Medication (Amiodarone) Post Surgical Ablation for Atrial Fibrillation - Is it Necessary?
Brief Title: Necessity of Anti-Arrhythmic Medication After Surgical Ablation for Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAM
Record Dates: First submitted 2011-03-21; First posted 2011-08-15 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Anti-Arrhythmic Medication
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Amiodarone (Active Comparator): Patient will be randomized not to receive to Amiodarone post Cox-Maze procedure unless indicated.
  Interventions: Other: No Amiodarone
- Amiodarone (No Intervention): Patients randomized to receive Amiodarone post Cox-Maze procedure which is our current standard of care.

INTERVENTIONS:
Other: No Amiodarone — This is a randomized study whereby patients who would routinely/usually be scheduled to receive Amiodarone as their anti-arrhythmic medication post surgical ablation will be randomly assigned to receive Amiodarone or no Amiodarone, but all other medications would remain as prescribed for patients following surgical ablation which will include beta blockade therapy unless contraindicated which is an American Heart Associated and Heart Rhythm Society recognized treatment.
  Arms: No Amiodarone

SUMMARY:
The purpose of this study is to determine whether anti arrhythmic medication, specifically Amiodarone, is required during the first three months post surgical ablation.

Hypothesis: Amiodarone will not be required during the first three months as verified by no increase in rehospitalizations for recurrent Atrial Fibrillation, and report of sinus rhythm at surgical follow up (approximately 3 weeks from date of surgery), 6 weeks and 12 weeks to include patients' first follow up with cardiologist at approximately 3 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject must be diagnosed with Persistent and/or Longstanding Persistent Atrial fibrillation as classified by the HRS Guidelines 8 [0]
* Subject must be selected as a candidate to undergo the Cox- Maze procedure for ablation of atrial fibrillation
* The Cox Maze procedure may be done as a stand alone procedure or combined with other cardiac surgical procedures either via a median sternotomy or a right thoracotomy:
* Subject has a Left Ventricular Ejection Fraction (LVEF) ≥ 30%
* Subject would normally be prescribed Amiodarone as an anti arrhythmic medication post surgical ablation
* Subject is able and willing to provide written informed consent and HIPAA authorization
* Subject is able and willing to comply with all study requirements including attending all follow-up visits as deemed necessary by personal physician (cardiologist)
* Subject has a life expectancy of at least one year

Exclusion Criteria:

* Subject has undergone previous attempts at surgical Maze procedure or other AF operation, including surgical or catheter ablation Subject has an accessory pathways disorder (e.g. Wolff-Parkinson-White syndrome)
* Subject is in Class IV NYHA
* Subject has had a documented MI within 6 weeks prior to study enrollment
* Subject needs emergent cardiac surgery (i.e. cardiogenic shock)
* Subject has known carotid artery stenosis greater than 80%
* Subject has a current diagnosis of active systemic infection
* Subject is pregnant, planning to become pregnant within 12-14 months, or lactating
* Subject requires preoperative intra-aortic balloon pump or intravenous inotropes
* Subject has renal failure requiring dialysis
* Subject is diagnosed with hepatic failure
* Subject is on anti-arrhythmic drug therapy for the treatment of a ventricular arrhythmia
* Subject has a known connective tissue disorder
* Subject is incarcerated
* Subject has previous or current therapy that could compromise tissue integrity including thoracic radiation, chemotherapy, long-term oral or injected steroids
* Subject is an intravenous drug and/or alcohol abuser
* Subject is participating in concomitant research studies of investigational products ( e.g. Appendage closure devices, atrial septal defect patches)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Status of Rhythm Between Baseline and Follow-Up - Recurrence of Atrial Fibrillation | 3, 6, 12 weeks and 6 months post-procedure
  To demonstrate equality in clinically significant recurrence of AF following ablation while showing superiority for complication and side effect rates in those off Amiodarone vs. those on.
  •% recurrence AF by telemetry at 3 wks and 24-48 hr Holter monitoring at 6 and 12 wks post procedure, EKG at first visit between 6 and 12 wks post discharge and or ER visit for rapid heart rate in atrial arrhythmia requiring treatment; permanent pacemaker interrogation reports at first follow up visit.
  •Post-procedure major adverse event rate at 6 mos post-procedure related to side effects of Amiodarone.

SECONDARY OUTCOMES:
Major Adverse Event Rate | 30 days post-procedure
  To characterize the composite post-procedure major adverse event rate (pericardial/ pleural effusion with elevated INR, hemorrhagic stroke with elevated INR, thromboembolic stroke) within 30 days post-procedure or prior to hospital discharge whatever comes last

CONTACTS AND LOCATIONS:
Overall Officials: Niv Ad, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

REFERENCES:
- [Derived] Ad N, Holmes SD, Shuman DJ, Pritchard G, Miller CE. Amiodarone after surgical ablation for atrial fibrillation: Is it really necessary? A prospective randomized controlled trial. J Thorac Cardiovasc Surg. 2016 Mar;151(3):798-803. doi: 10.1016/j.jtcvs.2015.07.034. Epub 2015 Jul 17. PMID 26253874